CLINICAL TRIAL: NCT01724905
Title: Weight Loss and Maintenance for Individuals With Intellectual Developmental Disabilities (IDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Donnelly (Other)
Responsible Party: Sponsor-Investigator, Joseph Donnelly, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18808
Record Dates: First submitted 2012-10-01; First posted 2012-11-12 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Weight Loss
Keywords: Diet; Obesity; Chronic disease
MeSH Terms: conditions — Weight Loss; Obesity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Stop Light Diet (Experimental)
  Interventions: Dietary Supplement: Modified Stop Light Diet (SLDm)
- Recommended Care for Weight Reduction (Active Comparator)
  Interventions: Dietary Supplement: Recommended Care Diet

INTERVENTIONS:
Dietary Supplement: Modified Stop Light Diet (SLDm) — SLDm includes reduced energy pre-packaged meals (PM) for 6 months, encouraged consumption of low energy shakes and 35 fruits and vegetables (F/V) per week
  Arms: Modified Stop Light Diet
Dietary Supplement: Recommended Care Diet — RC diet includes traditional meal plans and 35 fruits and vegetables per week
  Arms: Recommended Care for Weight Reduction

SUMMARY:
Individuals with intellectual developmental disabilities (IDD) have obesity rates that exceed those in the general population, consume energy dense diets, and perform very little physical activity (PA). Overweight and obesity are independent risk factors for chronic disease such as cancer, diabetes, hypertension, and cardiovascular disease in both the general population and those with IDD.

The investigators modified the Stop Light Diet (SLDm) to include reduced energy pre-packaged meals (PM) for 6 months, encouraged consumption of low energy shakes and 35 fruits and vegetables (F/V) per week. The investigators will compare participants who use the SLDm with participants who use a reduced energy and fat diet with meal plans, based off of the current American Dietetic Association recommended car for weight reduction plan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mile to moderate IDD as determined by a Community Service Provider operating in Kansas under the auspices of a Community Developmental Disability Organization (CDDO)
* Able to understand and give informed consent
* If there is a guardian with power of attorney, both the guardian and participant must give informed consent
* Participants must live in a supported living condition either at home or with no more than 1-4 residents and have a care giver (ie. parent, staff) who assists with food shopping, meal planning, and meal preparation
* Overweight or obese determined by a BMI > 25 kg/m2
* Able to walk
* Clearance provided from physician
* Able to communicate preferences

Exclusion Criteria:

* Uncontrolled hypertension
* Severe heart disease
* Cancer diagnosis
* Positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Weight loss between experimental diet (SLDm) and recommended care diet (RC) | Change from Baseline in Weight at 6 months
  The experimental diet is the Stop Light Diet modified (SLDm) and includes PM, 35 F/V per week, and low energy shakes. The Investigators will compare this to the RC diet that uses traditional meal plans and includes 35 F/V per week. Weight to be measured following an overnight fast of approximately 12 hours. Weight will be measured in kg. Each person will be weighed in a hospital gown between 8 and 10 am, using a calibrated scale to the nearest 0.1kg.
Weight loss between experimental diet (SLDm) and recommended care diet (RC) | Change from Baseline in Weight at 18 months
  The experimental diet is the Stop Light Diet modified (SLDm) and includes PM, 35 F/V per week, and low energy shakes. The Investigators will compare this to the RC diet that uses traditional meal plans and includes 35 F/V per week. Weight to be measured following an overnight fast of approximately 12 hours. Weight will be measured in kg. Each person will be weighed in a hospital gown between 8 and 10 am, using a calibrated scale to the nearest 0.1kg.

SECONDARY OUTCOMES:
Comparison of chronic disease factors - Blood Pressure | Change from Baseline in Blood Pressure at 18 months
  Changes in values of blood pressure between the two groups
Comparison of chronic disease factors - Glucose | Change from Baseline in Glucose at 18 months
  Changes in values of glucose between the two groups
Comparison of chronic disease factors - HDL | Change from Baseline in HDL-cholesterol Pressure at 18 months
  Changes in values of HDL-cholesterol between the two groups
Comparison of chronic disease factors - LDL | Change from Baseline in LDL-cholesterol Pressure at 18 months
  Changes in values of LDL-cholesterol between the two groups
Comparison of chronic disease factors - Insulin | Change from Baseline in Insulin Pressure at 18 months
  Changes in values of insulin between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Ptomey LT, Willis EA, Sherman JR, White DA, Donnelly JE. Exploring the effectiveness of an 18-month weight management intervention in adults with Down syndrome using propensity score matching. J Intellect Disabil Res. 2020 Mar;64(3):221-233. doi: 10.1111/jir.12713. Epub 2020 Jan 15. PMID 31944472
- [Derived] Ptomey LT, Steger FL, Lee J, Sullivan DK, Goetz JR, Honas JJ, Washburn RA, Gibson CA, Donnelly JE. Changes in Energy Intake and Diet Quality during an 18-Month Weight-Management Randomized Controlled Trial in Adults with Intellectual and Developmental Disabilities. J Acad Nutr Diet. 2018 Jun;118(6):1087-1096. doi: 10.1016/j.jand.2017.11.003. Epub 2018 Jan 6. PMID 29311038
- [Derived] Ptomey LT, Willis EA, Lee J, Washburn RA, Gibson CA, Honas JJ, Donnelly JE. The feasibility of using pedometers for self-report of steps and accelerometers for measuring physical activity in adults with intellectual and developmental disabilities across an 18-month intervention. J Intellect Disabil Res. 2017 Aug;61(8):792-801. doi: 10.1111/jir.12392. PMID 28707359